CLINICAL TRIAL: NCT07132242
Title: Safety and Efficacy of SHR-A1811 Combine With Pyrotinib for the Treatment of HER2 Positive Locally Advanced or Metastatic Breast Cancer, a Phase II Study
Brief Title: SHR-A1811 Combine With Pyrotinib for Locally Advanced/Metastatic HER2 Positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-092
Record Dates: First submitted 2025-08-01; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer With HER2 Positive
Keywords: SHR-A1811; Pyrotinib; HER2 positive; metastatic breast cancer; locally advanced breast cancer; Antibody drug conjugates
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1：SHR-A1811 4.0mg/kg + Pyrotinib 240mg/Day (Experimental)
  Interventions: Drug: SHR-A1811 4.0mg/kg; Drug: Pyrotinib 240mg
- Arm 2：SHR-A1811 4.0mg/kg + Pyrotinib 320mg/Day (Experimental)
  Interventions: Drug: SHR-A1811 4.0mg/kg; Drug: Pyrotinib 320mg
- Arm 3: SHR-A1811 4.8mg/kg + Pyrotinib 240mg/Day (Experimental)
  Interventions: Drug: Pyrotinib 240mg; Drug: SHR-A1811 4.8mg/kg
- Arm4: SHR-A1811 4.8mg/kg + Pyrotinib 320mg/Day (Experimental)
  Interventions: Drug: SHR-A1811 4.8mg/kg; Drug: Pyrotinib 320mg

INTERVENTIONS:
Drug: SHR-A1811 4.0mg/kg — SHR-A1811 4.0mg/kg, IV, Day 1, Q3W
  Arms: Arm 1：SHR-A1811 4.0mg/kg + Pyrotinib 240mg/Day; Arm 2：SHR-A1811 4.0mg/kg + Pyrotinib 320mg/Day
Drug: Pyrotinib 240mg — Pyrotinib 240mg, po, QD, from Day 8 to Day 21,Q3W
  Arms: Arm 1：SHR-A1811 4.0mg/kg + Pyrotinib 240mg/Day; Arm 3: SHR-A1811 4.8mg/kg + Pyrotinib 240mg/Day
Drug: SHR-A1811 4.8mg/kg — SHR-A1811 4.8mg/kg, IV, D1, Q3W
  Arms: Arm 3: SHR-A1811 4.8mg/kg + Pyrotinib 240mg/Day; Arm4: SHR-A1811 4.8mg/kg + Pyrotinib 320mg/Day
Drug: Pyrotinib 320mg — Pyrotinib 320mg, po, QD, from Day 8 to Day 21, Q3W
  Arms: Arm 2：SHR-A1811 4.0mg/kg + Pyrotinib 320mg/Day; Arm4: SHR-A1811 4.8mg/kg + Pyrotinib 320mg/Day

SUMMARY:
The goal of this clinical trial is to learn if SHR-A1811 combine with Pyrotinib is safe and tolerable for patients with HER2 positive breast cancer. It will also learn about the anti-tumor efficacy of this combination therapy. Participants will take SHR-A1811 and pyrotinib every three weeks, until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old and ≤70 years old;
* Pathologically confirmed HER2-positive locally advanced or metastatic breast cancer;
* Progression during or after prior HER2-targeted therapy and chemotherapy in the advanced/metastatic setting OR progression during/within 12 months after completion of trastuzumab and taxane-based chemotherapy in the neoadjuvant/adjuvant setting OR after 2 cycles of trastuzumab and taxane-based chemotherapy in the neoadjuvant setting with suboptimal response (assessed as non-response) for locally advanced disease;
* At least one measurable lesion per RECIST v1.1 criteria.
* ECOG performance status of 0 or 1.
* Adequate Organ Function
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose. Male subjects with partners of childbearing potential must be surgically sterile or agree to use effective contraception during the trial. Sperm donation is not permitted during the study period.
* Subjects must voluntarily enroll in this study, sign the informed consent form, demonstrate good compliance, and be willing to cooperate with follow-up.

Exclusion Criteria:

* Prior Pyrotinib in Advanced/Metastatic Setting;
* Prior Tropoisomerase I Inhibitor ADC Therapy;
* Active CNS Metastases;
* Other Malignancy;
* Recent Major Surgery/Trauma;
* Interstitial Lung Disease (ILD)/Severe Pulmonary Conditions;
* Significant Cardiac Disease;
* Inability to swallow oral medication, chronic diarrhea, intestinal obstruction, or other factors significantly affecting drug ingestion or absorption;
* Known hypersensitivity to any component of the investigational drugs in this study protocol;
* Immunodeficiency/Organ Transplant;
* Uncontrolled Third-Space Fluid Accumulation;
* Pregnancy/Breastfeeding/Contraception;
* Severe concomitant illness or comorbid conditions that may interfere with planned treatment or preclude study participation, as assessed by the investigator. This includes, but is not limited to, active hepatitis B or pulmonary infection requiring treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the date of signing ICF until the end of the safety follow-up period, defined as 40 days after the last administration of SHR-A1811 or Pyrotinib
  the proportion of patients who experienced treatment-emergent adverse events during the study treatment among the total number of patients experienced study treatment.
ORR | from initiation of the study treatment until disease progression (or treatment discontinuation), the observation period is up to 36 months.
  Objective Response Rate: The proportion of subjects achieving a best overall response(per RECIST v1.1) of complete response (CR) or partial response (PR) during the period from initiation of the study treatment until disease progression (or treatment discontinuation), relative to the total number of subjects in the analysis set.

SECONDARY OUTCOMES:
PFS | from the date of enrollment until the first documented radiological disease progression (PD) or death from any cause, the observation period is up to 36 months.
  progression free survival: the time interval from the date of ICF assigned until the first documented radiological disease progression (PD) or death from any cause. For subjects who had not experienced PD or death by the data cutoff date, or had received subsequent anti-cancer therapy, censoring will occur at the date of the last valid tumor assessment prior to the data cutoff date, or the initiation date of new anti-cancer therapy, whichever occurs first .
OS | The time from the date of enrollment to the date of death due to any cause. The observation period is up to 60 months.
  over all survival: The time from the date of enrollment to the date of death due to any cause. For subjects alive at the last follow-up , OS will be censored at the date of last contact . For subjects lost to follow-up , OS will be censored at the last date the subject was verified alive .Censored OS is defined as the time from enrollment to the censoring date.
DoR | from the date of first documented response to the date of disease progression or death of any cause, the observation period is up to 36 months.
  Duration of response:The time interval from the date of first documented response (complete response [CR] or partial response [PR], whichever is recorded earlier) until the date of disease progression or death of any cause.

IPD SHARING:
Plan to Share IPD: Undecided